## Statistical Analysis Plan

## Effects of Sleep hygiene Education on Sleep Health in Adults Ages 50 -80

Dr. Pfeiffer

Updated: 09/02/2024

NCT: 06129045

Approved by human subject protection review board committee on 09/02/2024

## Data Analysis

Statistical analyses will begin with the collection and reporting of demographic information for all study participants. This information will provide context for the sample and allow for appropriate interpretation of study outcomes.

Pre- and post-intervention survey data will be analyzed using paired-sample t tests. This approach will compare participant scores from the surveys administered at the beginning of the study to scores from the same surveys administered at the conclusion of the study, allowing for assessment of within-subject changes over time.

In addition to survey measures, objective sleep tracker data will be analyzed using paired-sample t tests. This will allow for comparison of baseline sleep measures with post-intervention measures, providing an additional source of quantitative evidence regarding the impact of the intervention.

All statistical analyses will be conducted using appropriate statistical software, and significance will be set at p < .05.